CLINICAL TRIAL: NCT01788956
Title: Correlation of Venous Oxygen Saturation Measurements by Non-invasive Mespere Venous Oximeter vs Central Venous Oxygen Saturation, Measured by a CO-Oximeter.
Brief Title: Comparison of Central Venous Oxygen Saturation Measurements by Non-invasive Mespere Venous Oximeter and Central Venous Catheter
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mespere Lifesciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MLS STP-9100002
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-09

CONDITIONS: Sepsis; Post Cardiac Surgery Low Output Syndrome Requiring Inotropic/Vasopressor Therapy; Cardiogenic Shock Post Myocardial Infarction; Hypoxemic Respiratory Failure.
Keywords: venous oximeter; CO-Oximeter; ICU Patients; Sepsis; non-invasive device
MeSH Terms: conditions — Sepsis; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU Patients: 80 subjects (male and female)
  Interventions: Device: Mespere Venous Oximeter; Device: Co-Oximeter

INTERVENTIONS:
Device: Mespere Venous Oximeter — Mespere Venous oximeter provides non-invasive measurement of the oxygenation of the venous blood.
Device: Co-Oximeter

SUMMARY:
The intent of this study is to validate the venous blood oxygenation measurements of the Mespere VA Oximeter compared to the saturations measured by venous blood sampling through an inserted central vein catheter, which is currently the standard of care for measuring SvO2

DETAILED DESCRIPTION:
The conventional bedside pulse oximeter has been a standard in clinical care for non-invasive hemodynamic monitoring and measures arterial blood oxygenation. To date, a non-invasive bedside monitor for measuring mixed venous oxygen saturation (SvO2) has not been developed. The clinical applications of venous oximetry are numerous and include management of severe sepsis and septic shock, trauma and hemorrhagic shock, heart failure and cardiac arrest.

The existing method for venous blood oxygenation monitored is either through an invasive fiber optic catheter, or intermittently by blood sampling through a central venous catheter Oximetry. However, SvO2 measurements using fiber optic catheters are very expensive, and all central line insertions include inherent risks. Also, insertion of a central line is in some circumstances not feasible (e.g. discomfort/limited experience in central line insertion, unavailability of specific monitoring systems etc.) resulting in inappropriate therapy usually guided by SvO2. Therefore, a non-invasive monitor to measure SvO2 at the bedside negating the requirement for a central line insertion would be of clinical benefit and allow appropriate therapy of many patients listed above at a time when therapy has the most benefit.

The Mespere VA Oximeter is a non-invasive medical device for monitoring of venous blood oxygenation.

Continuous measurement of venous oxygenation will be beneficial because it will help the physician better understand local ischemia as well as provide better guidance for the physician to be able to best treat the patient and decrease their burden of illness.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older
* Patients admitted to the ICU
* Patients who have or are scheduled to have an indwelling central venous catheter inserted via the internal jugular vein or subclavian vein as part of their usual care

Exclusion Criteria:

* Abnormal neck anatomy
* Unable to identify jugular vein under ultrasound guidance
* Allergic to adhesive tape
* Presence of known anatomical shunt or AV dialysis fistula
* Known central vein stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will consist of patients admitted either to the Medical Surgical ICU or the Cardiac Surgery Recovery Unit at University Hospital. The four groups will comprise patients with the following diagnoses: i) sepsis +/- septic shock, ii) post cardiac surgery low output syndrome requiring inotropic/vasopressor therapy, iii) cardiogenic shock post myocardial infarction, and iv) hypoxemic respiratory failure.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Mespere Venous Oximeter Accuracy Verification Study | up to 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Sharpe, MD, FRCPC, Principal Investigator — LHSC University Hospital
Locations (1):
- London Health Sciences Center, University Hospital, London, Ontario, Canada